CLINICAL TRIAL: NCT05947526
Title: Evaluation of the Outcomes of the Embryos Obtained From Different Follicle Sizes, and the miRNA Detection in the Spent Media of Their Blastocyst Culture
Brief Title: Outcomes of the Embryos of Different Ovarian Follicle Sizes, and the miRNA Detection in Their Blastocyst Culture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nazli Albayrak, Resident, MD, Acibadem University
Other Study IDs: 2023-10/349
Record Dates: First submitted 2022-11-23; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Embryo Quality
Keywords: follicle size; micro RNA; blastocyst culture; embryo quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women referring to infertility clinic for IVF treatment: Women who were referred to infertility clinic with complaint of not having baby go through IVF treatment, and having oocyte pick-up procedure with different sizes of ovarian follicles
  Interventions: Procedure: Oocyte pick-up

INTERVENTIONS:
Procedure: Oocyte pick-up — With the needle, transvaginally USG-guided oocyte pick-up procedure is going to be performed

SUMMARY:
In this study, it is aimed to analyze the outcomes of embryos obtained from ovarian follicle with different sizes, and identify the microRNA expression in the spent media of the blastocysts cultures.

DETAILED DESCRIPTION:
In this study, it is aimed to analyze the outcomes of embryos obtained from ovarian follicle with different sizes. By this way, we assume to predict which follicle is able to give the best blastocyst. After the blastocysts are obtained from the different sized follicles, blastocyst cultures are going to be studied for the up and down-regulations of microRNA, besides the correlation of embryo quality with miRNA expression in the spent media.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 20-38 who are planned to have IVF treatment
* On the day of trigger before the oocyte pick-up, patients having at least 5, and 14 at most follicles exceeding 11mm
* Patient having BMI below 30

Exclusion Criteria:

* PCO patients
* Patients having endometriosis
* Patients having male factor with severe oligoazoospermia

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients must be all female, since the study is based on embryos obtained from different ovarian follicle sizes
Study Population: Patients who are going to be included to the study will be the patients of infertility clinic
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Oocyte grading | after each hyper stimulation process of the patients, when the follicle sizes are large enough to pick up which is roughly 10-15 days after the hyper stimulation has started
  Morphologic Oocyte grading will be analyzed right after the procedure due to different follicle sizes
Day-3 Embryo Grading | Three days after the intracytoplasminc sperm injection(ICSI) procedure
  Morphologic Day-3 embryo grading will be analyzed after the procedure due to different follicle sizes
Day-5 Embryo Grading | 5 days after the intracytoplasminc sperm injection(ICSI) procedure
  Day-5 embryo grading(Gardner classification) will be analyzed after the procedure due to different follicle sizes
beta hCG results of the transferred embryos | ten days after the embryo transfer
  Clinical pregnancy outcomes

SECONDARY OUTCOMES:
micro RNA expression in culture medium | Culture mediums of day 5 embryos will be collected to be studied, after the last embryo is obtained and all will be studied at the end of the recruitment
  In the culture medium of blastocysts are going to be analyzed for microRNA levels that are expressed

CONTACTS AND LOCATIONS:
Overall Officials: NAZLI ALBAYRAK, MD, Principal Investigator — Acıbadem University School of Medicine
Locations (1):
- Acibadem University Atakent Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD is not going to be shared with other researchers. All data is going to be known only by one researcher.

REFERENCES:
- [Background] Shapiro BS, Rasouli MA, Verma K, Raman A, Garner FC, Aguirre M, Kaye L, Bedient C. The effect of ovarian follicle size on oocyte and embryology outcomes. Fertil Steril. 2022 Jun;117(6):1170-1176. doi: 10.1016/j.fertnstert.2022.02.017. Epub 2022 Mar 30. PMID 35367061
- [Background] Mohr-Sasson A, Orvieto R, Blumenfeld S, Axelrod M, Mor-Hadar D, Grin L, Aizer A, Haas J. The association between follicle size and oocyte development as a function of final follicular maturation triggering. Reprod Biomed Online. 2020 Jun;40(6):887-893. doi: 10.1016/j.rbmo.2020.02.005. Epub 2020 Feb 20. PMID 32389425
- [Background] Costermans NGJ, Soede NM, van Tricht F, Blokland M, Kemp B, Keijer J, Teerds KJ. Follicular fluid steroid profile in sows: relationship to follicle size and oocyte qualitydagger. Biol Reprod. 2020 Mar 13;102(3):740-749. doi: 10.1093/biolre/ioz217. PMID 31786607
- [Background] Rosen MP, Shen S, Dobson AT, Rinaudo PF, McCulloch CE, Cedars MI. A quantitative assessment of follicle size on oocyte developmental competence. Fertil Steril. 2008 Sep;90(3):684-90. doi: 10.1016/j.fertnstert.2007.02.011. Epub 2008 Feb 4. PMID 18249377
- [Background] Annes K, Muller DB, Vilela JAP, Valente RS, Caetano DP, Cibin FWS, Milazzotto MP, Mesquita FS, Belaz KRA, Eberlin MN, Sudano MJ. Influence of follicle size on bovine oocyte lipid composition, follicular metabolic and stress markers, embryo development and blastocyst lipid content. Reprod Fertil Dev. 2019 Mar;31(3):462-472. doi: 10.1071/RD18109. PMID 30282571
- [Background] Orvieto R, Mohr-Sasson A, Blumenfeld S, Nahum R, Aizer A, Haas J. Does a Large (>24 mm) Follicle Yield a Competent Oocyte/Embryo? Gynecol Obstet Invest. 2020;85(5):416-419. doi: 10.1159/000510876. Epub 2020 Sep 23. PMID 32966987
- [Background] Kasapoglu I, Orhan A, Aslan K, Sen E, Kaya A, Avci B, Uncu G. Are all antral follicles the same? Size of antral follicles as a key predictor for response to controlled ovarian stimulation. J Obstet Gynaecol. 2022 Apr;42(3):461-466. doi: 10.1080/01443615.2021.1910640. Epub 2021 Jun 22. PMID 34155958
- [Background] Saith RR, Srinivasan A, Michie D, Sargent IL. Relationships between the developmental potential of human in-vitro fertilization embryos and features describing the embryo, oocyte and follicle. Hum Reprod Update. 1998 Mar-Apr;4(2):121-34. doi: 10.1093/humupd/4.2.121. PMID 9683350
- [Background] Wittmaack FM, Kreger DO, Blasco L, Tureck RW, Mastroianni L Jr, Lessey BA. Effect of follicular size on oocyte retrieval, fertilization, cleavage, and embryo quality in in vitro fertilization cycles: a 6-year data collection. Fertil Steril. 1994 Dec;62(6):1205-10. doi: 10.1016/s0015-0282(16)57186-6. PMID 7957985
- [Background] Orvieto R, Mohr-Sasson A, Aizer A, Nahum R, Blumenfeld S, Kirshenbaum M, Haas J. Do Follicles of Obese Patients Yield Competent Oocytes/Embryos? Gynecol Obstet Invest. 2020;85(3):290-294. doi: 10.1159/000508226. Epub 2020 Jun 2. PMID 32485714